CLINICAL TRIAL: NCT00497107
Title: Phase III Randomized Controlled Clinical Study of UFT/LV Therapy Versus UFT/LV + PSK Therapy as Postoperative Adjuvant Therapy for Histological Stage IIIa and IIIb Colorectal Cancer
Brief Title: Uracil and Tegafur/Leucovorin (UFT/LV) Versus UFT/LV+ Polysaccharide-K (PSK) for Stage IIIa/IIIb Colorectal Cancer
Acronym: ICOG
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Iwate Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICOG-CC01
Record Dates: First submitted 2007-07-05; First posted 2007-07-06 (Estimated); Last update posted 2008-07-31 (Estimated); Status verified 2008-07

CONDITIONS: Colorectal Cancer
Keywords: UFT/LV; PSK; Colorectal cancer; Adjuvant therapy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Tegafur; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): The Control Group (UFT + Calcium Folinate)
  Interventions: Drug: UFT, Calcium Folinate
- 2 (Experimental): The PSK Group (UFT + Calcium Folinate + PSK)
  Interventions: Drug: UFT, Calcium Folinate, PSK

INTERVENTIONS:
Drug: UFT, Calcium Folinate, PSK
  Arms: 2
Drug: UFT, Calcium Folinate
  Arms: 1

SUMMARY:
The purpose of this study is to conduct a randomised controlled trial (RCT) comparing UFT/LV and UFT/LV + PSK in patients with histological stage IIIa/IIIb colorectal cancer who have undergone curative surgery without residual cancer using 3-year disease free survival (DFS) as the primary endpoint, and also to analyze the 3-year overall survival (OS), compliance, adverse events, quality of life (QOL) and relationship with tumor factors.

DETAILED DESCRIPTION:
To conduct a randomized controlled trial comparing chemotherapy using UFT/LV and immunochemotherapy using UFT/LV combined with PSK in patients with histological stage IIIa and IIIb colorectal cancer (adenocarcinoma) who have undergone curative surgery without residual cancer (R0) using 3-year disease-free survival rate as primary endpoint, and also to analyze the 3-year overall survival, compliance, adverse events, QOL and relationship with tumor factors.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a histological diagnosis of primary colon or rectal cancer (adenocarcinoma)
* Patient with histological stage IIIa or IIIb cancer (according to the Japanese Classification of Colorectal Cancer, 7th edition)
* Patient who has undergone curative surgery with no residual cancer
* Pretreatment criterion: patient who has not undergone preoperative cancer treatment (radiotherapy, chemotherapy or immunotherapy)
* Patient who is at least 20 years and below 80 years of age
* Patient with performance status (PS) of 0-1 (according to Eastern Cooperative Oncology Group, ECOG)
* Restrictions of concomitant medications and therapies: except in the case of metastasis or recurrence, concomitant use of other chemotherapeutic and immunotherapeutic agents that may affect the results of this trial, and concomitant use of radiotherapy are prohibited in principle.
* Organ function (laboratory data): patient who satisfies the following conditions or data of laboratory tests conducted within 2 weeks prior to start of trial

  * Gastrointestinal function: no diarrhea (watery stool)
  * White blood cell count: > 4,000/mm3
  * Platelet count: > 100,000/mm3
  * Serum GOT and GPT: < 100 IU/L
  * Serum total bilirubin: < 2.0 mg/dL
  * Serum creatinine: below the upper limit of facility normal range

Exclusion Criteria:

* Patient with residual cancer (R1 or R2)
* Patient with anal canal lesion (P) or perianal skin lesion (E)
* Patient with stricture and not capable of oral intake
* Patient passing fresh blood from the gastrointestinal tract
* Patient with retention of body cavity fluid necessitating treatment
* Patient with infection, intestinal palsy or intestinal occlusion
* Patient with active multiple cancers or patient who has less than 5 years of remission from a metachronous cancer (except carcinoma in situ and skin cancer)
* Patient who is pregnant or wishes to become pregnant during this trial
* Patient on continuous insulin treatment for diabetes or has poorly controlled diabetes
* Patient with a history of ischemic heart disease and judged to have difficulties to participate in this trial
* Patient with concurrent psychiatric disease or neurological symptoms and judged to have difficulties to participate in this trial
* Patient on continuous steroid therapy
* Patient with a history of serious drug allergy
* Patient who is judged for other reasons by the investigator or doctor in charge to be inappropriate as a subject

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2007-07; Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival | 3-years

SECONDARY OUTCOMES:
Overall survival, compliance, adverse events, QOL, tumor markers | 3-years

CONTACTS AND LOCATIONS:
Overall Officials: Go Wakabayashi, MD, PhD, Study Director — Iwate Clinical Oncology Group
Locations (1):
- Iwate Medical University Hospital, Morioka, Iwate, Japan

REFERENCES:
- [Background] Ohwada S, Ikeya T, Yokomori T, Kusaba T, Roppongi T, Takahashi T, Nakamura S, Kakinuma S, Iwazaki S, Ishikawa H, Kawate S, Nakajima T, Morishita Y. Adjuvant immunochemotherapy with oral Tegafur/Uracil plus PSK in patients with stage II or III colorectal cancer: a randomised controlled study. Br J Cancer. 2004 Mar 8;90(5):1003-10. doi: 10.1038/sj.bjc.6601619. PMID 14997197
- [Background] Lembersky BC, Wieand HS, Petrelli NJ, O'Connell MJ, Colangelo LH, Smith RE, Seay TE, Giguere JK, Marshall ME, Jacobs AD, Colman LK, Soran A, Yothers G, Wolmark N. Oral uracil and tegafur plus leucovorin compared with intravenous fluorouracil and leucovorin in stage II and III carcinoma of the colon: results from National Surgical Adjuvant Breast and Bowel Project Protocol C-06. J Clin Oncol. 2006 May 1;24(13):2059-64. doi: 10.1200/JCO.2005.04.7498. PMID 16648506